CLINICAL TRIAL: NCT06903221
Title: A Phase 4, Randomised Vaccination Study in Healthy Adults to Investigate the Effects of Acellular Pertussis Vaccine on Colonisation with Bordetella Pertussis Using Controlled Human Infection
Acronym: KIM
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dimitri Diavatopoulos (Other)
Responsible Party: Sponsor-Investigator, Dimitri Diavatopoulos, Senior researcher, Radboud University Medical Center
Organization: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023-508416-35-00; 2023-508416-35-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-02

CONDITIONS: Pertussis Infection; Pertussis Vaccines
Keywords: Controlled human infection model; Pertussis; Pertussis vaccine; Acellular pertussis vaccine; Tdap-IPV
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tdap-IPV - standard inoculum dose (Experimental): Participants get vaccinated with Tdap-IPV and will be challenged with 10E5 CFU Bordetella pertussis
  Interventions: Drug: Tdap-IPV
- Td-IPV - standard inoculum dose (Placebo Comparator): Participants get vaccinated with Td-IPV and will be challenged with 10E5 CFU Bordetella pertussis
  Interventions: Drug: Td-IPV
- Tdap-IPV - high inoculum dose (Experimental): Participants get vaccinated with Tdap-IPV and will be challenged with 10E6 CFU Bordetella pertussis
  Interventions: Drug: Tdap-IPV

INTERVENTIONS:
Drug: Tdap-IPV — intramuscular injection
  Other Names: acellular pertussis vaccine
  Arms: Tdap-IPV - high inoculum dose; Tdap-IPV - standard inoculum dose
Drug: Td-IPV — intramuscular injection
  Arms: Td-IPV - standard inoculum dose

SUMMARY:
The goal of this clinical trial is to investigate the effect of booster vaccination with acellular pertussis vaccine on colonization with Bordetella pertussis using a controlled human infection model in healthy volunteers. The main questions it aims to answer are:

* Whether booster vaccination with Tdap-IPV reduces Bp colonisation after intranasal challenge with the standard Bp inoculum dose compared to the Td-IPV control group
* Compare Bp colonisatation in participants vaccinated with Tdap-IPV after intranasal challenge with the standard and a 'high' Bp inoculum dose

Research will compare Tdap-IPV vaccination - standard inoculum dose with Td-IPV vaccination - standard inoculum dose, and Tdap-IPV vaccination - standard inoculum dose with Tdap-IPV vaccination - high inoculum dose to see how Tdap-IPV vaccination and the high inoculum dose have an effect on colonisation rate.

Participants will be vaccinated with Tdap-IPV or Td-IPV and 2-4 months later challenged with the standard or 'high' inoculum. After challenge there is a follow up visit for 28 days in which they fill in a daily symptom diary and have 6 visits to the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Participant (male/female) is born before 1-9-2004 and < 50 years old on the day of screening
* Participant has received all primary pertussis vaccines during childhood
* Participant is in good health as confirmed by review of medical history and physical examination
* Participant has adequate understanding of the procedures of the study and agrees to abide strictly thereby
* Participant is able to answer all questions of the pre-consent questionnaire correctly
* Participant is fully conversant in the Dutch language
* Participant is capable and willing to give personal signed informed consent.
* Participant is able to communicate by both mobile telephone and text messaging
* Participant is willing and available to attend all study visits
* Participant agrees to inform his/her general practitioner (GP) about participation in the study
* Participant agrees to provide access to information regarding their vaccination background
* Participant agrees to provide a treating physician access to all study-related information and data
* Participant is able to arrive within 1h at the Radboudumc from his/her home address. The participant must have a home address and live in the Netherlands
* Participant is able to arrive within 3h at the Radboudumc at any time between Bp inoculation until the day 28 post challenge visit
* Participant is willing to take an antibiotic regimen after inoculation with Bp according to the study protocol
* Participant is willing to use infection control measures during social contact during the study
* Participant is willing to attend to the Radboudumc immediately if they become symptomatic

Exclusion Criteria:

* Incapacitated subjects without decision-making capacity.
* A confirmed diagnosis of pertussis in the last two years and/or serum IgG anti-FHA >56 IU/mL
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (e.g., anaphylaxis) to any component of the study intervention.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Individuals who are at risk of complications of a prolonged cough, such as individuals with stress urine incontinence, pelvic floor dysfunction or an inguinal hernia
* Chronic use of i) immunosuppressive drugs (e.g. systemic steroids, steroid nasal spray or isotretinoin), ii) antibiotics, iii) or other immune modifying drugs within three months prior to study onset (topical corticosteroids and oral anti-histamines exempted) or expected use of such during the study period.
* Individuals with a history of autoimmune disease or an active autoimmune disease requiring therapeutic intervention.
* Drug or alcohol abuse interfering with normal social function in the period of one year prior to study onset
* Diabetes mellitus
* Smoking: Any smoking event in the last month, including (e-)cigarette, joint, cigar and pipe
* Infection with Bp or any other Bordetella species at the baseline for challenge visit
* Individuals who have a history of receiving pertussis vaccination in the last 5 years
* Acute illness within 3 days prior to Bp inoculation (including mild upper respiratory tract infection, common cold, running nose)
* Any antibiotic treatment within 4 weeks before inoculation
* Receipt of any non-study vaccine within 14 days, before and after receiving the study vaccine or Bp inoculation
* For female participants: pregnancy, lactation or intention to become pregnant during the study. Female volunteers are required to use an effective form of contraception during this study. Acceptable forms of contraception include:

  * Established use of oral, injected or implanted hormonal methods of contraception
  * Placement of an intrauterine device or intrauterine system
  * Total hysterectomy
  * Barrier methods of contraception (condom or occlusive cap with spermicide)
  * Male sterilisation if the vasectomised partner is the sole partner for the participant
  * True abstinence when this is in line with the preferred and usual lifestyle of the participant
* Known hypersensitivity to or contra-indications (including co-medication) for use of azithromycin or macrolides, see: azitromycine (oraal) (farmacotherapeutischkompas.nl). This includes: Clinically relevant bradycardia, hypokalemia, hypocalcemia and hypomagnesemia, cardiac arrhythmia or severe heart failure, congenital or acquired QT-prolongation, use of comedication which can cause QT-prolongation or is contraindicated co-medication: for a full list see: azitromycine (oraal) (farmacotherapeutischkompas.nl) - interactions.
* Participation in any other clinical study (unless observational) in the three months prior to the start of the study or during the study period
* Being an employee or student of the department of Laboratory Medicine, Radboudumc
* Any other condition or situation that would, in the opinion of the investigator, place the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol
* Individuals who have inviolable commitments within the study period during the challenge (28 days in total) to make contact with:

  * infants aged < 1 year
  * unimmunized children aged < 4 years
  * pregnant women >32 weeks who have not received pertussis vaccination at least a week prior to contact
  * chronically ill patients (e.g. asthma, COPD, heart diseases)
* Individuals who have household contacts working with

  * infants aged < 1 year
  * pregnant women
* The use of mouthwash during the challenge (35 days)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Bordetella pertussis (Bp) colonisation rate | Day 3-28 post challenge
  Bp colonisation rate in Tdap-IPV and Td-IPV vaccination groups, with Bp colonisation defined as any positive Bp culture from nasal wash samples at any time point between Day 3 and Day 28 after challenge

SECONDARY OUTCOMES:
Safety: solicited adverse events (AEs) | Day 0-28 post challenge
  Occurrence and intensity of respiratory and systemic symptoms of pertussis disease, from the challenge visit (V6) until day 28 after challenge (V12), per study group
Safety: azithromycin treatment | Day 0-28 post challenge
  Proportion of participants, per study group, that receive azithromycin treatment after Bp challenge (V6) and before day 28 (V12) as a result of development of early symptoms of pertussis disease
Safety: unsolicited AEs | Day 0-28 post challenge
  Occurrence and intensity of unsolicited adverse events, from the challenge visit (V6) until day 28 after challenge (V12), per study group
Colony forming unit (CFU) counts | Day 3-28 post challenge
  Bacterial load, defined as the number of colony forming units (CFUs) of Bp per ml detected in nasal wash of challenged participants at each sampling timepoint from day 3 (V7) until day 28 after challenge (V12), per study group
Geometric mean concentration of Bp-specific antibodies | 5 months
  Geometric mean concentration of Bp-specific antibodies in blood and mucosal samples at vaccination baseline (V2), 28 days post vaccination (V4), challenge baseline (V5) and 28 days post challenge (V12), per study group

CONTACTS AND LOCATIONS:
Locations (1):
- RadboudUMC, Nijmegen, Netherlands